CLINICAL TRIAL: NCT03316235
Title: New, Easy and Efficient Ways to CLassify AcetabulaR Fractures
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CLARIFY
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acetabular fractures are the resultant from high-energy trauma or low-energy trauma in the elder patients. Usually, surgeons use LETOURNEL's classification or/and JUDET's one.

Five elements are considered and associated to five type of fracture. Even more, for orthopaedic surgeons with less experience with these fractures, correct classification can be more difficult.

So the the aim of this study is:

1. Evaluate the efficacy of four "special" 3D reconstruction: a 3D reconstruction of the pelvis with anterior view, posterior view, endopelvic view where the opposite hemipelvis removed and an exopelvic view where the femoral head is removed according to the initial teaching of E. Letournel.
2. Evaluate the addition of teaching of non-experimented surgeon on the accuracy of classifying acetabular fractures.
3. Evaluate the addition of a digital algorithm (mobile application) on the accuracy of classifying acetabular fractures.

DETAILED DESCRIPTION:
12 reviewers will be given the different imaging of each case and will be divided in 4 groups: novice (junior ER and ortho residents), intermediate (non-experimented orthopedic surgeons), intermediate with a formation on classifying acetabular fractures and finally experts (acetabular fracture expert surgeons) . For each patient, representative CT scans are provided for each assessment. The study will be divided into 3 phases separated by 4-6 weeks of time. In the first phase, for each patient, representative CT scans are provided for each assessment with 2D and multiplanar reconstruction (MPR) without 3D views. In the second phase, 3D views are added. In the third phase, the cases are evaluated using the "Acetabular Diagnosis Tool" To note, the evaluation of the cases is done twice in each phase separated by 4-6 weeks and the order of the cases is changed, both in order to minimize recall bias

ELIGIBILITY:
Inclusion Criteria:

* acetabular fracture

Exclusion Criteria:

* no criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acetabular fracture surgery
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
3D reconstruction of pelvis CT scan | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France